CLINICAL TRIAL: NCT06280508
Title: A Prospective, Single-arm Exploratory Trail of Chemotherapy Combined With Adebrelimab and Apatinib as the Perioperative Treatment in Patients With Biliary Tract Cancer
Brief Title: Chemotherapy Combined With Adebrelimab and Apatinib as the Perioperative Treatment in Patients With Biliary Tract Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-082-01
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Resectable Intrahepatic Cholangiocarcinoma With High Risk of Recurrence
MeSH Terms: interventions — apatinib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental)
  Interventions: Drug: Adebrelimab, Apatinib, Gemcitabine, cisplatin

INTERVENTIONS:
Drug: Adebrelimab, Apatinib, Gemcitabine, cisplatin — Chemotherapy combined with Adebrelimab and Apatinib neoadjuvant therapy for 3 cycles before surgery, and Adebrelimab combined with Apatinib adjuvant therapy for 6 months after surgery

SUMMARY:
This is a prospective, single-arm exploratory study to evaluate the efficacy and safety of chemotherapy combined with Adebrelimab and Apatinib as the perioperative treatment in Patients With Biliary Tract Cancer.

ELIGIBILITY:
Inclusion Criteria:

* confirmed intrahepatic cholangiocarcinoma
* with Resectable tumor lesion
* no contraindications to surgery
* with high risk of tumour recurrence
* No prior systemic therapy for intrahepatic cholangiocarcinoma.
* ECOG Performance Status of 0 or 1
* Child-Pugh Class: Grade A

Exclusion Criteria:

* History of gastrointestinal hemorrhage within 6 months prior to the start of study treatment or clear tendency of gastrointestinal hemorrhage
* Abdominal fistula, gastrointestinal perforation or intraperitoneal abscess within 6 months prior to the start of study treatment
* Known genetic or acquired hemorrhage or thrombotic tendency
* Thrombosis or thromboembolic event within 6 months prior to the start of study treatment
* Cardiac clinical symptom or disease that is not well controlled
* Hypertension that can not be well controlled through antihypertensive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
1-year EFS rate | Up to approximately 3 years
  1-year event-free survival rate

SECONDARY OUTCOMES:
R0 Resection rate | Up to approximately 3 years
  R0 Resection rate
EFS | Up to approximately 3 years
  Event-free survival
RFS | Up to approximately 3 years
  Recurrence-free survival
OS | Up to approximately 3 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yajin Chen, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, China/Guangdong, China

IPD SHARING:
Plan to Share IPD: No